CLINICAL TRIAL: NCT01527422
Title: Protocol CCAM 05-02 " Phase I-II Study of Dose Dense of PEG Filgrastim and GM-CSF as Support for Dose Desnse CHOP-R Front Line Therapy for Aggressive Non Hodgkin's Lymphoma"
Brief Title: Cyclophosphamide, Doxorubicin, Vincristine, Prednisone, Rituximab Pateinets With Aggresive NHL
Acronym: CHOP-R
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fernando Cabanillas (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Fernando Cabanillas, Hematolgy-Oncologyst, Auxilio Mutuo Cancer Center
Organization: Auxilio Mutuo Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT01297478; NCT01297478 (obsolete NCT alias)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma; Non Hodgkin's Lymphoma
Keywords: Aggressive Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Rituximab; Granulocyte Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cyclophosphamide, Doxorubicin, Vincristine and Prednisone — Rituximab will be administered on day 1 of courses 1-6 at 375 mg/m2 concurrently with CHOP-R.All patients will receive antiemetics priorchemotherapy.Courses will be repeated every 14 days.If blood counts don't allow re-treatment on day 14 the counts will be repeated at least twice per week until recovery allows re-treatment.The aim is to achieve a dose that will be as close as possible to 250 mcg and that will result in grade 0 or grade 1A or 1B toxicity at the most. The dose of PEG-Filgrastim will initially be fixed at 3 mg until dose level +3 is reached (which includes 250 mcg Leukine) at which time the dose of Neulasta will be escalated if necessary. All patients will receive Neulasta as a subcutaneous injection on the day 3.
  Other Names: Cyclophosphamide (Cytoxan); Doxorubicin (Adryamicin); Vincristine (Oncovin); Prednisone; Rituximab (Rituxan); Peg Filgrastim[Neulasta (G-CSF or GCSF)]; Leukine (Sargramostim)

SUMMARY:
We now propose to investigate the combination of CHOP-Rituxan plus PEG-Filgrastim (PEG-filgrastim) and GM-CSF. PEG-Filgrastim would be given in order to allow us to administer the chemotherapy courses every 2 weeks with the practical advantage of requiring only one dose of PEG-filgrastim instead of daily doses of G-CSF.

DETAILED DESCRIPTION:
1.1 Primary Objective:

1. To identify the ideal dose of the combination of CHOP-R with PEG-Filgrastim (Neulasta) using first a fixed dose of Neulasta and an escalating dose of GM-CSF (Leukine) up to 250 mcg. When that dose is reached, if possible, the dose of Neulasta will be increased stepwise. CHOP-R will be delivered every 14 days at a fixed standard dose with dose adjustments of PEG-Filgrastim and GM-CSF upwards and downwards according to nadir or zenith blood counts.

   1.2 Secondary Objective:
2. To generate preliminary pilot data as to the effectiveness of the regimen in inducing very early remissions as measured by the CT-PET scan technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated aggressive non-Hodgkin's Lymphoma. Aggressive histologies include follicular large cell, diffuse large cell, peripheral T cell, transformed lymphomas, Lymphoblastic lymphomas, Burkitt and Burkitt like lymphomas.
* Must have measurable or evaluable disease.
* Stage I-IV patients are eligible
* Patients must be 18 years or older.
* No evidence of grade 3 or more neurosensory or neuromotor dysfunction (see appendix- toxicity criteria)
* Written Consent

Exclusion Criteria:

* HIV positive patients and those with Hepatitis B or C will be excluded from this protocol.
* Patients with inadequate bone marrow and organ function as defined below:
* Neutrophils <1,000/l
* Platelets <100,000/l
* Billirubin >2
* Creatinine >2.0 or estimated CrCl <30 cc/min
* CNS involvement by Lymphoma.
* Uncontrolled intercurrent disease including arrhythmias, angina pectoris, Class III-IV Congestive heart failure (CHF symptoms on less than ordinary exertion or at rest) or active infection.
* Active infection or fever > 38.2 degrees C unless due to lymphoma.
* Subject is not using adequate contraceptive precautions.
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Phase I-II Study of Dose Dense of PEG-Filgrastim and GM-CSF combined with CHOP-R | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Auxilio; Fernando Cabanillas, MD, Principal Investigator — Auxilio Mutuo Cancer Center/Hospital Auxilio Mutuo
Locations (1):
- Hospital Auxilio Mutuo Cancer Center, San Juan, Puerto Rico, Puerto Rico